CLINICAL TRIAL: NCT06992323
Title: Cardiometabolic Properties of Omega-3 Funcionalized With Hydroxytyrosol in Healthy and Cardiovascular Risk Population
Brief Title: Cardiometabolic Properties of Omega-3 Functionalized With Hydroxytyrosol
Acronym: HydroxyOmega
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Council, Spain (Other Government)
Collaborators: Beps Holding GmbH (Unknown); Olivenova Health Sl (Unknown)
Responsible Party: Principal Investigator, María Raquel Mateos Briz, Principal Investigator, National Research Council, Spain
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: HYDROXYOMEGA
Record Dates: First submitted 2025-04-10; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-04

CONDITIONS: Hypertriglyceridemia; Normal
Keywords: cardiovascular risk; omega 3; hydroxytyrosol; hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia | interventions — Sunflower Oil

STUDY DESIGN:
Intervention Model Description: Chronic, randomized, controlled, cross-over, double-blind, and free-living study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- EPA + HT (Experimental): EPA + HT: intake of 2 g/d of EPA and 15 mg/d of HT (3 Type-1 capsules, EPA + HT)
  Interventions: Dietary Supplement: EPA + HT
- EPA (Experimental): EPA: intake of 2 g/d of EPA (3 Type-2 capsules, EPA)
  Interventions: Dietary Supplement: EPA
- Sunflower oil (SO) (Active Comparator): Sunflower Oil (SO): intake of 2 g/d of SO (3 Type-3 capsules, Placebo)
  Interventions: Dietary Supplement: Sunflower Oil

INTERVENTIONS:
Dietary Supplement: EPA + HT — Volunteers will consume during 12 weeks 2 g/d of EPA and 15 mg/d of HT, corresponding to 3 capsules. Additionally, they will consume a commercial olive oil with a minimal phenol content as their culinary oil that will be suplied by the research team for family use (1L/2 weeks)
  Arms: EPA + HT
Dietary Supplement: EPA — Volunteers will consume during 12 weeks 2 g/d of EPA corresponding to 3 capsules. Additionally, they will consume a commercial olive oil with a minimal phenol content as their culinary oil that will be suplied by the research team for family use (1L/2 weeks)
  Arms: EPA
Dietary Supplement: Sunflower Oil — Volunteers will consume during 12 weeks 2 g/d of Sunflower Oil, corresponding to 3 capsules. Additionally, they will consume a commercial olive oil with a minimal phenol content as their culinary oil that will be suplied by the research team for family use (1L/2 weeks)
  Arms: Sunflower oil (SO)

SUMMARY:
The primary aim of this study is to investigate the potential cardioprotective effects of daily nutritional doses of eicosapentaenoic acid (EPA) enriched with hydroxytyrosol (HT) on cardiovascular health, as well as its modulatory impact on the intestinal microbiota. This investigation will be conducted through a randomized, double-blind, crossover, and controlled nutritional intervention trial. The study population will include two cohorts: one with normotriglyceridemic individuals, and another with hypertriglyceridemic individuals. Participants will be randomly allocated to one of three intervention groups: (1) EPA+HT supplementation, (2) EPA alone, or (3) a placebo consisting of sunflower oil devoid of EPA.

DETAILED DESCRIPTION:
The product to be tested is a combination of two key components: an oily preparation containing 97% eicosapentaenoic acid (EPA) and a natural extract (Oleacore®) with a high hydroxytyrosol content (10%). Oleacore® is naturally derived from olives using exclusively physical and mechanical methods and is commercialized by Olivenova Health SL (https://olivenova.com/es/). The EPA-97% component is supplied by Beeps Holding GMBH (https://bepsholding.com/el-holding/?lang=es). Three types of nutraceutical formulations will be prepared, and study participants will consume three capsules daily to achieve the following dosages:

1. 2 g of EPA + 15 mg of hydroxytyrosol (HT) (3 Type-1 capsules, EPA+HT),
2. 2 g of EPA (3 Type-2 capsules, EPA), and
3. 2 g of seed oil (sunflower) as a placebo (3 Type-3 capsules, Placebo).

The daily dose of 15 mg HT was selected based on the EFSA claim for the prevention of LDL oxidation , while the 2 g EPA dose was established following EFSA recommendations for triglyceride reduction.

A chronic, randomized, controlled, crossover, double-blind, free-living study design is proposed, spanning 46 weeks. Following a two-week washout period, during which the consumption of extra virgin olive oil, and olives will be restricted, participants will be grouped based on baseline characteristics (control or hypertriglyceridemia). They will then be randomized into three groups (randomization performed using SPSS software), such that one-third of participants will receive EPA+HT, another third will receive EPA without HT, and the remaining third will receive a placebo nutraceutical containing sunflower oil with no EPA or HT.

Each intervention phase will last 12 weeks. After completing one intervention, participants will undergo a four-week washout period before transitioning to the next intervention. Before the start of each phase, participants will be provided with all necessary capsules (EPA+HT, EPA, or placebo) along with detailed consumption guidelines.Volunteers will take the capsules with lunch and dinner.

Additionally, during the study, volunteers will consume a commercial olive oil with a minimal phenol content as their culinary oil. This olive oil will also be supplied by the research team for family use (1 L/2 weeks). Participants will be instructed to maintain their usual lifestyle throughout the study but will be restricted from consuming any other culinary oils apart from the one provided by the research group, as well as olives. Furthermore, the use of dietary supplements containing antioxidants, other than vitamins, will be prohibited.

Participants will attend the Human Nutrition Unit (UNH) at ICTAN-CSIC on six occasions, corresponding to the beginning and end of each intervention phase. Once eligibility has been confirmed based on the inclusion and exclusion criteria, participants will attend the UNH for signing the informed consent, receiving olive oil for household consumption, and receiving instructions to begin the study.

During visits V1-V6 (corresponding to the start and end of each intervention with the different nutraceuticals), participants will report to the UNH at ICTAN-CSIC. Upon arrival, they will provide a fasting urine sample from their first morning void and a stool sample collected within the previous 24 hours. Additionally, a trained nurse will collect a fasting blood sample (40 mL, distributed into tubes containing various anticoagulants).

Blood pressure and heart rate will also be measured. Furthermore, participants will undergo a comprehensive anthropometric and body composition assessment. Dietary habits and physical activity levels will be monitored and evaluated during these visits.

Compliance with the intervention will be monitored through monthly telephone follow-ups, the collection of unused capsules, and the measurement of specific biomarkers, including plasma phosphatidylcholine-EPA levels as a marker of omega-3 fatty acid intake and urinary HT metabolites.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 70 years old
* Hypertriglyceridemia (150-250 mg/dl) or normal levels of triglycerides levels (<150 mg/dl)

Exclusion Criteria:

* Presence of chronic illnesses
* Currently undergoing pharmacological treatment
* Smoking
* Pregnancy
* Adherence to a vegetarian or vegan diet

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Total cholesterol concentration | 12 months
  Total cholesterol in serum samples will be determined following reference methods recommended by the Sociedad Española de Bioquímica Clínica y Patología Molecular (SEQC) using the Roche Cobas Integra 400 plus analyser (Roche Diagnostics).
HDL-C, LDL-C, VLDL-C, and triglyceride concentrations | 12 months
  Measured in serum using reference or enzymatic methods recommended by SEQC.
Apolipoprotein A1 and B concentrations | 12 months
  Measured with clinical chemistry methods based on SEQC guidelines.
Aminotransferases: AST (ASAT) and ALT (ALAT) enzyme activity | 12 months
  Measured using enzymatic methods.
Uric acid, creatinine and glucose concentrations | 12 months
  Measured using standardised spectrophotometric methods.
Endothelial biomarkers | 12 months
  VCAM-1, ICAM-1, eNOS, E-selectin, and P-selectin concentrations will be measured in serum using ELISA.
Platelet function markers | 12 months
  Leukotriene B4 and prostaglandin E2 will be measured in serum using ELISAs (Cayman kits).
Serum cytokines (IL-6, IFN-γ, TNF-α, IL-10) | 12 months
  Serum concentrations of interleukin-6 (IL-6), interferon gamma (IFN-γ), tumor necrosis factor alpha (TNF-α), and interleukin-10 (IL-10) will be determined using ELISA. These biomarkers reflect both pro- and anti-inflammatory responses.
C-Reactive Protein (CRP) | 12 months
  CRP will be measured using an automated ultrasensitive turbidimetric method (AU2700 Biochemistry analyser, Olympus).
Oxidized LDL and 8-hydroxy-2'-deoxyguanosine (8-OHdG) | 12 months
  LDLox and 8-OHdG will be measured in serum using ELISA.
Lipid peroxidation (TBARS) | 12 months
  TBARS will be measured as µM MDA equivalents using ELISA.
TAS will be assessed using a colorimetric assay or ELISA. | 12 months
  TAS will be assessed using a colorimetric assay or ELISA.
Total oxidative status (TOS) | 12 months
  TOS will be measured using ELISA.
Antioxidant enzyme activities (NOX, GSH, GPx, SOD) | 12 months
  NADPH oxidase (NOX), glutathione (GSH), glutathione peroxidase (GPx), and superoxide dismutase (SOD) will be measured using ELISA-based methods.

SECONDARY OUTCOMES:
Systolic and Diastolic Blood Pressure | 12 months
  Systolic and diastolic blood pressure will be measured using an automatic arm sphygmomanometer (BS 150; Pic Indolor Diagnostic) at baseline and at the end of each intervention period. Measurements will be taken after the volunteer has rested on a chair for 5 minutes. Two consecutive readings will be taken on the left arm. If the values differ by more than 10-15 mmHg, a third reading will be recorded. The mean of the two (or three) closest readings will be used for analysis. Blood pressure will be expressed in mmHg..
Resting Heart Rate | 12 months
  Heart rate will be measured using the same automatic arm sphygmomanometer (BS 150; Pic Indolor Diagnostic) under the same conditions as blood pressure. Volunteers will rest for 5 minutes prior to the measurement. If multiple readings are required due to variation, the mean of the two (or three) closest values will be used. Heart rate will be expressed in beats per minute (bpm).
Fecal Short Chain Fatty Acids (SCFAs) Concentration | 12 months
  Short chain fatty acids (SCFAs) determination in faeces.The analytes will be analysed by gas chromatography system (Agilent Technologies Palo Alto, CA, USA) equipped with a mass spectrometer (MS) detector and Agilent DB-WAXtr column (100% polyethilen glycol, 60 m, 0.325 mm, 0250 um).
Fecal Lactate Concentration | 12 months
  Lactate levels in fecal samples will be measured using an Advanced Compact Ion Chromatographic instrument IC867 (Metrohm AG, Herisau, Switzerland).
Gut Microbiota Composition (16S rRNA Gene Profiling) | 12 months
  Microbial composition of fecal samples will be assessed by 16S rRNA gene amplicon sequencing. Genomic DNA will be extracted using the Quick-DNA™ Fecal/Soil Microbe Miniprep Kit (Zymo Research). Library preparation and sequencing will be conducted at Maastricht University (the Netherlands). Data analysis will be performed using the QIIME software package (v1.9.0), with taxonomic assignment based on the Greengenes database (v13.8).
Fasting glucose | 12 months
  Measured using SEQC-recommended methods.
Fasting insulin and C-peptide | 12 months
  Measured using immunoassays or ELISA.
Glycated hemoglobin (HbA1c) | 12 months
  Measured using HPLC or immunoturbidimetric methods.
Incretins (Glucagon and GLP-1) | 12 months
  Glucagon and GLP-1 concentrations will be measured using ELISA.
Adipokines (Leptin and PAI-1) | 12 months
  Leptin and plasminogen activator inhibitor-1 (PAI-1) will be measured using ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Mateos Briz Tenured Scientist, Principal Investigator — National Research Council (CSIC)
Locations (1):
- Institute of Food Science, Food Technology and Nutrition (ICTAN), CSIC, Madrid, Madrid, Spain